CLINICAL TRIAL: NCT05273463
Title: Comparison of Perioperative Education Modalities for ACL Reconstruction on Patient Satisfaction, Self-Efficacy, and Surgical Outcomes: A Randomized Controlled Trial
Brief Title: Comparing Perioperative Education Modalities for ACL Reconstruction on Patient Satisfaction, Self-Efficacy, and Surgical Outcomes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Hayley R. Powell, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-002443
Record Dates: First submitted 2022-02-24; First posted 2022-03-10 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: ACL Injury; Anterior Cruciate Ligament Injuries
Keywords: ACL Reconstruction
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Video-Based Education Group (Experimental): Approximately 4 weeks before scheduled surgery, participants will receive the video-based intervention regarding pre-and postoperative care for ACL reconstruction.
  Interventions: Behavioral: Video-Based Intervention
- Virtual Classroom Course Group (Experimental): Approximately 4 weeks before scheduled surgery, participants will receive the classroom-based intervention regarding pre-and postoperative care for ACL reconstruction.
  Interventions: Behavioral: Classroom-Based Intervention
- Standard of Care Group (No Intervention): Participants will receive verbal and written pre-and postoperative instruction as typically received by all ACL reconstruction patients treated by the attending physicians before and after surgery.

INTERVENTIONS:
Behavioral: Video-Based Intervention — 15-minute video about what to expect before, during, and after your surgery
  Arms: Video-Based Education Group
Behavioral: Classroom-Based Intervention — Virtual 30-minute course with an Orthopedic nurse about what to expect before, during, and after your surgery
  Arms: Virtual Classroom Course Group

SUMMARY:
The purpose of this research is to find out whether the way information about surgery is presented to patients affects patient satisfaction, knowledge retention, and surgical outcomes such as anxiety

ELIGIBILITY:
Inclusion Criteria:

* Patients of Senior Attending orthopedic sports medicine surgeons at Mayo Clinic Arizona
* Patients with a proficiency in English in order to participate without need for translator.
* Patients with a diagnosis of a primary ACL injury in need of surgical reconstruction utilizing any surgical technique for ACL reconstruction.

Exclusion Criteria:

* Patients with a diagnosis of ACL injury in need of a surgical revision.
* Patients who have any multi-ligamentous injuries to the knee requiring modified postoperative unloading.
* Patients who have history of previous anterior cruciate ligament reconstructions in either leg.
* Patients who have either auditory or visual impairments.
* Patients who are medical professionals with work-related knowledge of ACL reconstruction.
* Patients with an inability or unwillingness of individual or legal guardian to give written informed consent.

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2022-08-23 (Actual); Primary Completion 2025-12-02 (Actual); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Patient Satisfaction | 24 months
  Measured using the Leiden Perioperative Patient Satisfaction Questionnaire. Self-reported questionnaire that rates the subjects satisfaction with information provision, discomfort and needs during perioperative care.

SECONDARY OUTCOMES:
Anxiety | 24 months
  Measured using the PROMIS Emotional Distress - Anxiety Short Form 8a. Self-reported 8-item questionnaire that rates the subjects emotional distress in the past 7 days on a scale of 1=Never to 5=Always. Higher total scores indicate higher anxiety severity.
Self-Efficacy | 24 months
  Measured using the PROMIS Self-Efficacy - Manage Symptoms Short Form 8a. Self-reported 8-item questionnaire that rates the subjects current level of confidence to statements about managing symptoms using a scale of 1="I am not at all confident to 5="I am very confident". Higher total score indicate higher confidence in managing symptoms.
Kinesiophobia | 24 months
  Measured using the Tampa Scale for Kinesiophobia. Self-reported 17-item questionnaire based on evaluation of fear of movement, fear of physical activity, and fear avoidance using a scale of 1=Strongly Disagree to 4=Strongly Agree. Total score range from 17-68 and higher scores indicate severe kinesiophobia.
Physical Function | 24 months
  Measured using the PROMIS Physical Function Short Form 10b. Self-reported 10-item questionnaire that rates the subjects ability to perform an activity using a scale of 5="Without any difficulty" to 1="Unable to do". Higher total scores indicate higher physical function.
Knowledge Retention | 24 months
  Measured using the ACL Reconstruction Perioperative Education Quiz
Pain Interference | 24 months
  Measured using the PROMIS Pain Interference Short Form 6a. Self-reported 6-item questionnaire that rates the subjects pain interference with activities in the past 7 days using a scale of 1="Not at all" to 5="Very much". Higher total scores indicate higher pain interference with activities experienced.
History of Falls | 24 months
  Measured using the History of Falls Questionnaire. Self-reported 5-item questionnaire asking subjects about falls experienced in the past month and seriousness.
Lysholm Knee Score | 24 months
  Measured using the Lysholm Knee Scoring Scale. Self-reported questionnaire that asks subjects to indicate which statement best describes their condition in regards to common complaints frequently experience with knee problems. Total scoring out of 100 and higher score less knee-specific symptoms.
Activity Level | 24 months
  Measured using the Tegner Activity Scale. Self-reported level of activity prior to injury and post injury. Total of 10 levels and higher levels indicate greater activity level.
Confidence in Returning to Sport | 24 months
  Measured using the ACL Return to Sport Index. Self-reported 6-item questionnaire to measure the readiness to return to sports after ACL injury or reconstruction. Using a scale from 0 points (extremely negative psychological responses) to 100 points (no negative psychological responses).
Resilience | 24 months
  Measured using the Brief Resilience Scale. Self-reported 6-item questionnaire to measure perceived ability to recover from stress. Total score range 1-5 with higher scores indicating higher resilience.

CONTACTS AND LOCATIONS:
Overall Officials: Hayley Powell, MSN, RN, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Arizona, Phoenix, Arizona, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials